CLINICAL TRIAL: NCT07020247
Title: Personalized Long-course Radiotherapy Plus Chemotherapy With or Without Immunotherapy for Locally Advanced Rectal Cancer：A Randomized Controlled Study (PALACE Study)
Brief Title: Personalized Long-course Radiotherapy Plus Chemotherapy With or Without Immunotherapy for LARC: PALACE Study
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Wang Xin, Professor, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PALACE
Record Dates: First submitted 2025-04-06; First posted 2025-06-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2024-12

CONDITIONS: Locally Advanced Rectal Cancer (LARC); Immunotherapy; Radiotherapy; Total Neoadjuvant Therapy; Anal Function Preservation
MeSH Terms: interventions — Radiotherapy; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Total Neoadjuvant Chemoradiotherapy+Serplulimab (Experimental): The experimental group intervention consists of the following:
  1. Induction Phase: Two cycles of CAPOX and serplulimab prior to radiotherapy.
  2. Concurrent Chemoradiotherapy: Two cycles of CAPOX and serplulimab administered concurrently with radiotherapy.
  3. Consolidation Phase: Two additional cycles of CAPOX and serplulimab, initiated 2-3 weeks after completing radiotherapy.
  Radiotherapy is delivered using intensity-modulated radiotherapy (IMRT/VMAT) at a dose of 50-50.4Gy/25-28f (1.8-2.0Gy/d, 5f/w). For patients in the experimental group who achieve partial remission (PR) or better during the induction phase, an additional local boost dose of 6Gy/3f (2.0Gy/d, 5f/w) is administered to the PGTV.
  Tumor response is assessed 3-4 weeks after completing consolidation chemotherapy. Based on the evaluation, a decision is made to proceed with either total mesorectal excision (TME) or a watchful waiting strategy.
  Interventions: Drug: Anti-PD-1 antibody drug named Serplulimab; Radiation: Radiotherapy; Drug: Chemotherapy
- Total Neoadjuvant Chemoradiotherapy (Active Comparator): The control group intervention consists of the following:
  1. Induction Phase: Two cycles of CAPOX prior to radiotherapy.
  2. Concurrent Chemoradiotherapy: Two cycles of CAPOX administered concurrently with radiotherapy.
  3. Consolidation Phase: Two additional cycles of CAPOX, initiated 2-3 weeks after completing radiotherapy.
  Radiotherapy is delivered using intensity-modulated radiotherapy (IMRT/VMAT) at a dose of 50-50.4Gy/25-28f (1.8-2.0Gy/d, 5f/w).
  Tumor response is assessed 3-4 weeks after completing consolidation chemotherapy. Based on the evaluation, a decision is made to proceed with either total mesorectal excision (TME) or a watchful waiting strategy.
  Interventions: Radiation: Radiotherapy; Drug: Chemotherapy

INTERVENTIONS:
Drug: Anti-PD-1 antibody drug named Serplulimab — Serplulimab
  Arms: Total Neoadjuvant Chemoradiotherapy+Serplulimab
Radiation: Radiotherapy — Radiotherapy is delivered using intensity-modulated radiotherapy (IMRT/VMAT) at a dose of 50-50.4Gy/ 25-28f(1.8-2.0Gy/d, 5f/w). For patients in the experimental group who achieve partial remission (PR) or better during the induction phase, an additional local boost dose of 6Gy/3f(2.0Gy/d, 5f/w) is administered to the PGTV.(No PGTV dose was given in the control group). For the treatment of lymph node metastasis in the lateral pelvic wall outside the mesorectal area: no additional dose is required when surgery is feasible, a sequential boost dose of 15Gy/3f is added when the lymph nodes are not surgically resectable.
Drug: Chemotherapy — Capox

SUMMARY:
The study is a multicenter, randomized controlled, phase III clinical study, and the purpose of the study is to explore the complete response rate (CR, Defined as pathological complete response (pCR) + Clinical complete response (cCR) sustained for over one year) of patients with locally advanced rectal cancer(LARC) treated with personalized long-course radiotherapy plus chemotherapy with or without Serplulimab. A total of 184 patients were included in this study.

DETAILED DESCRIPTION:
Patients diagnosed with locally advanced rectal cancer (T3-4/N+) and presenting with combined risk factors, where the lower boundary of the lesion is ≤ 10 cm from the anal margin, will undergo neoadjuvant therapy. The primary endpoint of the study is the complete response rate (CR), defined as the combination of pathological complete response (pCR) and clinical complete response (cCR) sustained for over one year.

ELIGIBILITY:
Inclusion Criteria:

1. Age: ≥18 years old; sex is not limited.
2. Patients with stage II/III rectal cancer staged under MRI or endoscopic ultrasonography and have at least one risk factor: cT4a and invasion of intestinal lumen for more than 1/2 week (measured by MRI)；cT4b(resectable)；cT3c-d with EMVI+ (upper middle rectum)；cN2；MRF+ (≤2mm)；lower rectal cancer is located on the anterior wall and tumor reaching T3 and occupying the intestinal cavity for more than 1/2 week; lower rectal cancer is mainly located on the lateral posterior wall need invading the intestinal wall (anal sphincter) ≥ 5mm； tumor of lower rectal cancer invades the external anal sphincter or levator ani muscle (stage 4) . [According to the 8th edition of the 2018 AJCC Cancer Staging Manual and the 2008 ESMO Lower Segment Colorectal Cancer Staging Criteria] . The preoperative T stage is referred to endoscopic ultrasonography or rectal MRI. The N stage is referred to abdominal CT. The M stage is referred to abdominal and thoracic CT. If symptoms occur, other appropriate imaging examinations are needed (cranial MRI or ECT) . Patients with contraindications to MRI can be interpreted with caution based on CT and endoluminal ultrasound staging. MDT should review the staging of all patients.
3. The lower edge of lesion is less than 10cm from anal verge according to rigid sigmoidoscopy or rectal digital examination.
4. No distant metastasis after a thorough examination .
5. Pathological diagnosis of rectal adenocarcinoma,and Immunohistochemistry and/or genetic testing for MSS/pMMR;
6. ECOG score: 0-1.
7. Patients with primary rectal cancer who had not received surgery prior to surgery (except for palliative ileostomy or colostomy), radiotherapy, systemic chemotherapy or other anti-tumor therapy.
8. The main organ function is normal, including the following characteristics:

   ①Blood routine examination: HB ≥9g/dL, WBC ≥ 3.5/4.0×109/L，NE≥ 1.5×109/L，PLT≥ 100×109/L

   ②Biochemical examination：Crea and BIL ≤ 1.0 upper normal limit（ULN），ALT and AST≤ 2.5 upper normal limit（ULN）, ALP≤2.5×UNL，Tbil≤1.5×UNL。
9. Not allergic to 5-Fu or Platinum.
10. The site of radiotherapy had not previously received radiation.
11. If female and of childbearing potential, have a negative result on a pregnancy test performed a maximum of 7 days before initiation of study treatment. If female and of childbearing potential, or if male, agree to use adequate contraception (eg, abstinence, intrauterine device, oral contraceptive, or double-barrier method) based on the judgment of the investigator or a designated associate from the date on which the ICF (Informed Consent Form) is signed until 8 weeks after the last dose of study drug.
12. Participants are volunteered to participate in this study, sign informed consent, good compliance, cooperation with follow-up.

Exclusion Criteria:

1. Patients who have previously received pelvic radiotherapy.
2. Presence of active or progressive infection requiring systemic treatment, such as active tuberculosis, active hepatitis, etc.
3. Presence of systemic diseases that are not stably controlled by the investigator, including diabetes mellitus, hypertension, liver cirrhosis, rheumatic immune diseases, and severe lung diseases.
4. Have had prior or concurrent cancer distinct in primary site or histology (including synchronous colon cancer) , except for curatively treated cervical cancer in situ, Basal cell carcinoma of skin.
5. Has any other disease, metabolic abnormality, physical examination abnormality, or laboratory abnormality that, in the judgment of the investigator, has reason to suspect that the patient has a disease or condition for which the study drug is inappropriate for use, or that would affect the interpretation of the study results, or place the patient in a high-risk condition.
6. Estimated inadequate patient compliance to participate in this clinical study.
7. History of gastrointestinal fistula, perforation, bleeding or severe ulceration or presence of severe gastrointestinal disease that affects the absorption of oral chemotherapy drugs.
8. Patients who have received solid organ transplantation or bone marrow transplantation, or have had active autoimmune disease requiring systemic therapy within 2 years prior to the first dose.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Estimated)
Dates: Start 2024-11-19 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Complete response rate | 1 year
  Defined as the combination of pathological complete response (pCR) and clinical complete response (cCR) sustained for over one year.

SECONDARY OUTCOMES:
R0 resection rates | 1 year
  The proportion of patients achieved a complete resection with negative margin
Disease free survival | 3 years
  Time from the completion of the treatment to any recurrences or distant metastases
Anus-preserving rate | 1 year
  The rate of anal organ preservation patients to all patients
Locoregional recurrence-free survival (LRFS) rates | 3 years
  The rate of patients without local recurrence to all the patients
Distant metastasis free survival | 3 years
  Time from the completion of the treatment to any distant metastases
Overall survival | 3 years
  OS is defined as the difference between the date of study enrollment to the date death due to any cause
The adverse effects during the chemoradiotherapy | 3 months
  Any side effects during the chemoradiotherapy
Quality of life (QoL) | 1 year
  Assessed using the Chinese version of QLQ-C30 to measure quality of life
Surgical Safety Metrics | 1 year
  Surgical safety was assessed using the Clavien-Dindo classification system

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No